CLINICAL TRIAL: NCT03212573
Title: Impact of Implementation of an Enhanced Recovery After Surgery Program in Laparoscopic Roux-en-Y Gastric Bypass
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Research Department, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HRJC17/18
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Nurse evaluating postoperative pain is blinded to the protocol applied
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS protocol (Experimental): ERAS protocol includes early oral intake (6 hours after surgery), early deambulation (6h after surgery) and multimodal analgesia (port-sites infiltration with Bupivacain 0.5% combined with postoperative intravenous analgesia)
  Interventions: Combination Product: ERAS protocol
- Standard care (Active Comparator): Oral intake and early deambulation begins 24h after surgery and analgesia consists in only intravenous drugs
  Interventions: Combination Product: Standard care

INTERVENTIONS:
Combination Product: ERAS protocol — ERAS protocol includes early oral intake and deambulation and multimodal analgesia
  Arms: ERAS protocol
Combination Product: Standard care — Oral intake and deambulation 24h after surgery and only intravenous analgesia.
  Arms: Standard care

SUMMARY:
A prospective randomized study of patients undergoing Roux-en-Y gastric bypass will be randomized in 2 groups: those following an ERAS program and those ones following a standard protocol.

Postoperative pain 24 hours after surgery and hospital stay will be assessed.

DETAILED DESCRIPTION:
A prospective randomized study of patients undergoing Roux-en-Y gastric bypass will be randomized in 2 groups: those following an Enhanced Recovery After Surgery (ERAS) program and those ones following a standard protocol. The ERAS program implies early liquids oral intake, early deambulation and multimodal analgesia (port sites infiltration with Bupivacain 0.5% associated with intravenous analgesia).

Postoperative pain 24 hours after surgery, as measured by Visual Analogic Scale, and hospital stay will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >40 Kg/m2
* BMI >35 Kg/m2 with obesity-associated comorbidities

Exclusion Criteria:

* Patients undergoing other bariatric procedures
* Patients undergoing bariatric revisional surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after surgery
  Evaluated by Visual Analogic Scale

SECONDARY OUTCOMES:
Hospital stay | Days until patients´discharge: 2 days or more than 2 days
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Duran, Study Chair — Hospital Rey Juan carlos
Locations (1):
- General Hospital Elche, Elche, Alicante, Spain